CLINICAL TRIAL: NCT01580176
Title: A Prospective Clinical Trial on Agreement to Evaluate the GlucoseMonitor, a Novel Device for Continuous Assessment of Blood Glucose Levels, in Comparison With the RAPIDLab® 1265 Blood Gas Analyser (ContAssGlu)
Brief Title: Continuous GlucoseMonitor for Measurement of Blood Glucose Level
Acronym: ContAssGlu
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Susanne Frankenhauser (Other)
Responsible Party: Sponsor-Investigator, Susanne Frankenhauser, Dr. Susanne Frankenhauser, University Hospital Heidelberg
Organization: University Hospital Heidelberg (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: ContAssGlu
Record Dates: First submitted 2012-04-17; First posted 2012-04-18 (Estimated); Last update posted 2013-12-20 (Estimated); Status verified 2013-12

CONDITIONS: Other Surgical Procedures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GlucoseMonitor (Experimental)
  Interventions: Device: continuous GlucoseMonitor

INTERVENTIONS:
Device: continuous GlucoseMonitor — The blood glucose and blood lactate levels will be taken continuously by the Continuous GlucoseMonitor and will be recorded twelve times.
  Other Names: blood glucose examination stand

SUMMARY:
This study will be the first study in which the new central venous microdialysis-based continuous glucose monitoring system (Continuous GlucoseMonitor) is used to investigate the performance of this Continuous GlucoseMonitor, as the measurements will be compared with a point of care reference (RAPIDLab® 1265 blood gas analyser). Further important points are also much less blood samplings / blood loss for the patient and personnel costs.

DETAILED DESCRIPTION:
The current standard for measuring blood glucose concentrations on ICU is to manually draw a blood sample from an arterial catheter and analyse the sample using a point of care blood gas analyser. This technique has several disadvantages as causes considerable blood loss and does not produce a continuous blood glucose profile and it is labour intensive (multiple samples over time are needed to follow the changes in blood glucose concentration). The monitoring system (Continuous GlucoseMonitor) based on the microdialysis technique has the advantage that not blood, but a physiological fluid such as saline is used as test medium. In brief, a physiological fluid, called the perfusate is continuously perfused through the microdialysis probe. At the membrane of the probe, glucose (as other low-molecular weight molecules) diffuses from the surrounding sample into the perfusate, now called dialysate, and is transported outside the probe for ex vivo monitoring.

ELIGIBILITY:
Inclusion Criteria:

* having undergone major abdominal and predominantly pancreatic surgery due to any reason
* expected to be in intensive care for at least 8 hours following index surgery
* need for close monitoring of blood glucose levels postoperatively
* having received a two-lumen central venous catheter for anaesthesia and operative purposes
* antibiotic prophylaxis (e.g. mezlocillin 4.0g and metronidazole 500mg)
* received routine perioperative thromboembolic prophylaxis medication (e.g. low-molecular-weight-heparin, heparin)
* aged at least 18 up to 80 years
* Capable of giving informed consent (written informed consent, signed and dated)
* successful central venous catheter in place (at least double lumen)
* one lumen of the central venous catheter will not be used postoperatively for routine infusion therapy and routine application of medications

Exclusion Criteria:

* known history of thrombosis, embolism; vascular obliteration
* known bleeding disorders, e.g. thrombocytosis
* known history of acute or chronic renal failure and patients on renal replacement therapy (dialysis, hemofiltration)
* known history of acute or chronic heart failure
* evidence of acute postoperative hyperhydration (pulmonary congestion)
* known history of acquired immune deficiency syndrome
* patients receiving immune suppressive therapy
* any signs for acute or chronic infection
* contraindication for insertion of a central venous catheter
* contraindication for perioperative thromboembolic prophylaxis medication (e.g. low-molecular-weight-heparin, heparin)
* exceedance the flushing infusion volume (500 mL per 24 hours)
* pregnancy and lactation
* Participation in another parallel clinical trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-03; Primary Completion 2012-12 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Eight hours measurement after initial referencing | eight hours after initial referencing
  Agreement at point of care, i.e. agreement between the readings from the Continuous GlucoseMonitor taken eight hours after initial referencing and the measurement results from the RAPIDLab® 1265 blood gas analyser taken at the same time

SECONDARY OUTCOMES:
one and two (short) and three to eight (mid) deterioration | one, two, three, four, five, six, seven and eight hours
  Short (one and two hour) and mid term (three to eight hour) deterioration in agreement, i.e. agreement between the readings from the Continuous GlucoseMonitor taken one and two and three, four, five, six, seven as well as eight hours after initial referencing and the measurement results from the RAPIDLab® 1265 blood gas analyser taken at the same time

CONTACTS AND LOCATIONS:
Overall Officials: Johann Motsch, Prof. Dr., Principal Investigator — University Hospital Heidelberg, Department of Anaesthesiology
Locations (1):
- University Hospital Heidelberg, Department of Anaesthesiology, Heidelberg, Germany

REFERENCES:
- [Derived] Zimmermann JB, Lehmann M, Hofer S, Husing J, Alles C, Werner J, Stiller J, Kunnecke W, Luntz S, Motsch J, Weigand MA. Design of a prospective clinical study on the agreement between the Continuous GlucoseMonitor, a novel device for CONTinuous ASSessment of blood GLUcose levels, and the RAPIDLab(R) 1265 blood gas analyser: The CONTASSGLU study. BMC Anesthesiol. 2012 Sep 22;12:24. doi: 10.1186/1471-2253-12-24. PMID 22998112